CLINICAL TRIAL: NCT06692842
Title: Implementation Study of an Interactive Technological Intervention to Improve Mental Health Symptoms in Primary Health Care Users
Brief Title: Interactive Technological Intervention to Improve Mental Health Symptoms in Primary Health Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80837624.7.0000.0068
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Depression; Anxiety; Insomnia
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Individuals with anxiety, depression or insomnia will receive the CONEMO intervention, consisting of 7 self-applied modules of strategies based on cognitive-behavioral therapy techniques. The intervention will be comparet to the treatment as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONEMO (Experimental): CONEMO is a low-intensity psychoeducational program which is made available to users via smartphones compatible with Android or iOS systems. At the same time, the designed healthcare professional use a tablet to monitor user adherence to the intervention. CONEMO comprise seven weekly modules, totally self-guides.
  Interventions: Device: CONEMO App

INTERVENTIONS:
Device: CONEMO App — The CONEMO application has three protocol, aimed to improived symptoms of depression, insomnia and anxiety. It is based on cognitive behavioral therapy (CBT) and contextual behavioral therapy (activation behavioral theraphy, mindfulness) and adapted considering broader contexts of mental health care, which involves a low-intensity intervention administered without any or minimal professional guidance and widely accessible. In a brief and structured format, CONEMO involves offering the intervention through texts, audios and videos. Based on the principles of CBT and contextual thrapies, CONEMO is organized into structured sessions that promote psychoeducation and teach basic behavioral skills, often through interactive exercises. Each journey was developed based on scientific evidences. The CONEMO journeys comprise seven weekly modules.

SUMMARY:
This study aims to implement and evaluate a technological intervention called CONEMO to treat depressive symptoms, anxiety, and insomnia in adults who use primary health care services. The effectiveness of this intervention has already been proven in previous research, specifically for depressive symptoms. Implementation will occur in 28 basic health units in the municipalities of Indiatuba and Jaguariúna in the interior of São Paulo.

All eligible residents of the cities will be invited to participate.

DETAILED DESCRIPTION:
A type III hybrid implementation and effectiveness study, with a mixed-method explanatory sequential design consisting of two distinct stages: the first quantitative, followed by qualitative. The method is indicated when the researcher wishes to use qualitative data to help interpret and explain the initial quantitative findings and deepen them. The elements of both methods are analyzed separately and then merged, looking for convergences, divergences, contradictions, or relationships between the two databases.

The qualitative data will help to interpret, explain and deepen the quantitative findings. The guidelines of the Consolidated Criteria for Reporting Qualitative Research (COREQ) will be followed, a 32-item instrument that guides the conduct of the interview and analysis of qualitative data, also validated in Portuguese in Brazil.

Study site The study will be carried out in 28 Basic Health Units (UBS) in two municipalities in the interior of São Paulo, Indaiatuba and Jaguariúna, located approximately 100 km from the capital São Paulo, in the state of São Paulo, Brazil.

Study population - stakeholder groups Patients/service users - user category Our study population will be made up of adult individuals (18 years or older) who live in the municipality of Indaiatuba or Jaguariúna and attend the UBS and who show significant symptoms of depression, anxiety or insomnia.

Health professionals, service managers and local managers - professional categories Adults (18 years or older) from the groups of interest will also participate in the study: health professionals from the UBS in the municipalities of Jaguariúna and Indaiatuba, service managers, health department managers, or primary care and mental health coordinators. We consider these individuals to be the main stakeholders, in addition to the users and main participants in the research, in the unfolding of the CONEMO intervention implementation study.

Study population

User participants - quantitative study:

All individuals screened at the cities' UBSs with positive symptoms for insomnia, anxiety or depression.

Participants - users, health professionals and managers - barriers and facilitators - qualitative study The focus groups in this study will be divided into categories of participants selected from each UBS involved. The categories of participation will be users, technical health professionals, senior health professionals and the manager of each participating unit. Simple randomization will be carried out to select one participant from each category among users and health professionals. With regard to managers, the invitation will be extended to all managers of the participating health units. These focus groups will be conducted separately for each category of participants at the end of three months from the start of the study. It is important to note that the users included in the focus groups may be at different stages of using the application. Specific guiding scripts will be used to collect the qualitative data, which will be drawn up after analyzing the quantitative data.

Research Steering Committee - CGP This committee plays a crucial role in monitoring and evaluating the outcomes of the implementation of interventions and policies. Composed of a multidisciplinary team, including academic researchers, local managers, and service workers, the committee facilitates the active participation of all stakeholders in the research process. Its main objective is to ensure that contextual elements are taken into account and that real conditions are understood and worked on. The committee meets regularly to discuss the research progress, evaluate the strategies' implementation and provide constructive feedback. This participatory and collaborative approach helps to identify and overcome possible challenges in implementation, thus promoting the effectiveness and sustainability of the mental health policies implemented. The CGP will also include users of municipal health services.

ELIGIBILITY:
Inclusion Criteria:

* Look for consultation in basic health units due to Major Depressive Disorder, Insomnia and/or Generalized Anxiety Disorder, or who receive home visits for the same reason.
* Score >= 10 on the PHQ-9 Scale for Depression; and/or >= 11 on the IGI Scale for Insomnia; and/or >= 10 on the GAD-7 Scale for Anxiety.
* Be able to read the app's instructions via a tablet or smartphone screen.

Exclusion Criteria:

* Individuals considered severe on the Suicide Risk Assessment Protocol-SRAP (suicidal imminence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — the individual will declare the gender with which they identify
Enrollment: 12400 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who have 'recovered' from depressive symptoms (PHQ-9 < 10) | 3 months
  Patient Health Questionnaire-9 (PHQ-9) is a questionnaire to access the severity of participants' depressive symptoms. The PHQ-9 score varies according to the severity of the symptoms and is classified as follows: no depression (0 to 4), mild symptoms (5 to 9), moderate symptoms (10 to 14), moderately severe symptoms (15 to 19) and severe symptoms (20 to 27). A cut-off point of 10 is suggested to indicate the presence of significant depressive symptoms.
Proportion of participants who have 'recovered' from anxiety (GAD-7< 10) | 3 months
  General Anxiety Disorder-7 (GAD-7) scale, which measures common symptoms associated with generalized anxiety disorder in the last two weeks. Each of the scale's seven items ranges from 0 ('not at all') to 3 ('almost every day'), resulting in a total score ranging from 0 to 21. A suggested cut-off point of more than 10 points indicates the presence of anxiety.
Proportion of participants who have 'recovered' from insomnia (IGI<8) | 3 months
  Insomnia Severity Index (IGI) is a retrospective instrument that assesses the last month and is made up of seven items that explore various aspects of sleep, including difficulties initiating or maintaining sleep, early morning awakening, satisfaction with sleep, daytime impairment, perception of sleep problems by other people, and concern about sleep problems.
  Respondents use a Likert scale ranging from 0 (no severity) to 4 (high severity), resulting in a total score ranging from 0 to 28. This score is classified as follows: no insomnia (0 to 7), mild insomnia (8 to 14), moderate insomnia (15 to 21) and severe insomnia (22 to 28

SECONDARY OUTCOMES:
Social Support Assessment: | 3 months and 6 months
  The participant's relationships with other people, i.e. whether they have a support network, will be explored throught a questionnaire
Quality of Life | 3 months and 6 months
  The level 3 version of the 5-item EUROQol questionnaire (EQ 5D-3L), which covers five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with three levels of severity, will be used to access changes in quality of life.
Daily Activity Level: | 3 months and 6 months
  Through the short form of the Behavioral Activation Scale for Depression (BADS). The BADS is a 9-item scale that measures the frequency of activation and avoidance behaviors that are hypothetically fundamental to the mechanisms of depression. This instrument will only be applied to participants in the depression journey.

CONTACTS AND LOCATIONS:
Locations (1):
- Basic Health System, Indaiatuba and Jaguariúna, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared on the OSF platform after the study is completed, upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion and publication of the results
Access Criteria: Upon request from others researchers